CLINICAL TRIAL: NCT06932250
Title: Vascular and Neural Mechanisms of Chronic Leg Heating in Pregnant Women With Obesity
Brief Title: Leg Heating in Pregnant Women With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Qi Fu, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU20250500
Record Dates: First submitted 2025-03-19; First posted 2025-04-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: High-risk Pregnancy
Keywords: Pregnancy; Obesity; Heat therapy; Vascular function; Sympathetic neural control; Blood pressure
MeSH Terms: conditions — Obesity; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sauna blanket set at 65°C (Experimental): The temperature of the sauna blanket will be set at 65°C and participants will perform home-based leg heating 4 times per week, 45 minutes per session.
  Interventions: Other: Leg heating
- Sauna blanket set at 35°C (Placebo Comparator): The temperature of the sauna blanket will be set at 35°C and participants will perform home-based leg heating 4 times per week, 45 minutes per session.
  Interventions: Other: Leg heating

INTERVENTIONS:
Other: Leg heating — Participants will perform home-based leg heating using a portable sauna blanket set at different temperature.

SUMMARY:
Obesity is a major risk factor for hypertensive disorders of pregnancy (HDP). The underlying mechanisms are largely unclear, but maternal vascular endothelial dysfunction is likely involved. Endothelial dysfunction in HDP could be attributed to 1) alterations in the L-arginine/nitric oxide (NO) pathway, and 2) an increase in endothelin-1 (ET-1). Additionally, augmented sympathetic vasoconstriction may also contribute to HDP. Chronic (repeated) whole-body heat exposure has been shown to increase NO bioavailability, decrease ET-1, and cause functional and structural adaptations in the vasculature. All these can improve vascular function, attenuate sympathetic (re)activity, lower blood pressure (BP), and reduce cardiovascular risk in non-pregnant individuals. Whether this is also true after regional (leg) heating in high-risk pregnant women is unknown. The investigators' central hypothesis is that chronic leg heating will be effective in improving vascular endothelial function and attenuating sympathetic vasoconstriction, leading to a reduction of the risk for HDP in pregnant women with obesity. The overarching goal of this proposal is to determine the vascular and neural effects of chronic leg heating in obese pregnancy. The study team plans to enroll pregnant women with obesity between 12-14 weeks of gestation and randomly assign them to either an intervention group or a control group (1:1 ratio). Participants in the intervention group will perform 16 weeks of home-based leg heating using a portable sauna blanket up to the hip (temperature of the blanket will be set at 65°C, 4 times/week, 45 min/session), whereas women in the control group will set the temperature of the blanket at 35°C at the same frequency and duration. Participants will be evaluated at baseline and then at 28-30 weeks of gestation. Aim 1 will determine the effects of chronic leg heating on maternal vascular function and surrogate markers of HDP. Aim 2 will determine the effects of chronic leg heating on sympathetic vasoconstriction and BP. Findings from this project will provide insight on the extent and potential mechanisms of how chronic leg heating works for improving vascular endothelial function and sympathetic vasoconstriction in pregnant women with obesity. Results obtained will set a foundation for future large multicenter clinical trials to determine the efficacy and generalizability of home-based leg heat therapy as a safe, ease-of-use, cost-effective, and non-drug approach for reducing the risk of HDP.

DETAILED DESCRIPTION:
Obesity is a major risk factor for hypertensive disorders of pregnancy (HDP). The underlying mechanisms are unclear, but maternal vascular endothelial dysfunction is likely involved. Endothelial dysfunction in HDP could be attributed in part to: 1) alterations in the L-arginine/nitric oxide (NO) pathway, and 2) an increase in endothelin-1 (ET-1). Conversely, augmented sympathetic vasoconstriction may also contribute to the development of HDP in women with obesity. Exercise training increases NO production, decreases ET-1, improves vascular function, attenuates sympathetic (re)activity, and reduces the risk for HDP. However, pregnant women, especially those with obesity, have poor adherence to exercise. Thus, there is an urgent need to develop novel, safe, convenient, low-cost, and well-tolerated strategies that have similar beneficial effects as exercise training. One such novel approach may be "heating".

During passive whole-body heating, body core temperature increases and cutaneous and muscle vascular resistance decreases, leading to increases in blood flow and shear stress throughout the entire arterial tree. Chronic (i.e., repeated) exposure to these temperature-dependent responses induces an increase in NO bioavailability, a decrease in ET-1, and functional and structural adaptations in the vasculature - all these can improve vascular function, attenuate sympathetic (re)activity, lower blood pressure (BP), and reduce the risk for cardiovascular morbidity and mortality. Evidence suggests that maternal body core temperature below 38.9°C is safe for the fetus.

The study team proposes to use regional (e.g., leg) rather than whole-body (e.g., hot tub or sauna) heating, since leg heating does not substantially elevate body core temperature (i.e., 37.32°C at peak in pregnant women with obesity in our pilot study), is more tolerable than whole-body heating, and can be performed in-home. Importantly, the study team's preliminary work showed that chronic home-based leg heating is safe, and can improve endothelial function, attenuate sympathetic vasoconstriction, and reduce ambulatory awake BP in pregnant women with obesity.

The investigators' central hypothesis is that chronic leg heating will be effective in improving vascular endothelial function and attenuating sympathetic vasoconstriction, leading to a reduction of the risk for HDP in pregnant women with obesity.

Aim 1: Determine the effects of chronic leg heating on maternal vascular function and surrogate markers of HDP.

Hypothesis 1: Chronic leg heating will improve vascular endothelial function due to an increase in NO bioavailability and a decrease in ET-1, which may be associated with a reduction of the risk for HDP in pregnant women with obesity.

Aim 2: Determine the effects of chronic leg heating on sympathetic vasoconstriction and BP.

Hypothesis 2: Chronic leg heating will attenuate sympathetic-dependent vasoconstriction due to a decrease in sympathetic (re)activity, which may be associated with a reduction of BP in pregnant women with obesity.

Impact: Findings from this project will provide insight on the extent and potential mechanisms of how chronic leg heating works for improving vascular endothelial function and sympathetic vasoconstriction in pregnant women with obesity. Results obtained will set a foundation for future large multicenter clinical trials to determine the efficacy and generalizability of home-based leg heat therapy as a safe, ease-of-use, cost-effective, and non-drug approach for reducing the risk of HDP, and its most severe form, preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women with overweight or obesity (self-reported pre-pregnancy body mass index ≥25 kg/m2) between 10-14 weeks of gestation and aged 18-45 years old will be enrolled.
* Both normotensive and hypertensive (office sitting systolic BP 140-150 mmHg and/or diastolic BP 90-100 mmHg) pregnant women will be enrolled if they are not on any antihypertensive drug treatment.
* We will enroll both nulliparous and multiparous women.
* There is no restriction regarding race/ethnicity and socioeconomic status.
* Women with a history of HDP will be allowed to participate.
* Women taking low-dose aspirin will be allowed to participate and aspirin use will be documented.

Exclusion Criteria:

* Current multiple pregnancies (e.g., twins, triplets, etc.).
* Known major fetal chromosomal or anatomical abnormalities diagnosed during the study.
* Recurrent miscarriage (three or more, to avoid antiphospholipid antibody syndrome).
* Office sitting BP <100/55 mmHg or >150/100 mmHg (for safety reasons).
* Evidence of cardiovascular, pulmonary, or neurological diseases.
* Diabetes mellitus (to avoid its effects on vascular endothelial function and sympathetic vasoconstriction).
* Kidney disease (serum creatinine >0.9 mg/dL).
* Clinical known deep vein thrombosis, clinical symptoms and history of deep vein thrombosis, or dermatological lesions.
* History of drug or alcohol abuse within the last 2 years.
* Current tobacco use.
* Pregnant women who do not have air conditioning at home during summer (for safety reasons).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in vascular endothelial function | Baseline, 16 weeks after leg heating
  Change in vascular endothelial function assessed by brachial artery flow-mediated vasodilation using the Doppler ultrasound technique
Change in sympathetic neural control | Baseline, 16 weeks after leg heating
  Change in sympathetic neural control assessed by muscle sympathetic nerve (re)activity using the microneurographic technique
Change in sympathetic vascular transduction | Baseline, 16 weeks after leg heating
  Change in sympathetic vascular transduction assessed using the microneurographic and Doppler ultrasound techniques

SECONDARY OUTCOMES:
Change in blood concentration of nitrate | Baseline, 16 weeks after leg heating
  Blood concentration of nitrate will be used to estimate nitric oxide bioavailability
Change in blood concentration of nitrite | Baseline, 16 weeks after leg heating
  Blood concentration of nitrite will be used to estimate nitric oxide bioavailability
Change in L-arginine level | Baseline, 16 weeks after leg heating
Change in asymmetric dimethylarginine level | Baseline, 16 weeks after leg heating
Change in 3-nitrotyrosine level | Baseline, 16 weeks after leg heating
Change in concentration of endothelin-1 | Baseline, 16 weeks after leg heating
Change in 24-hour ambulatory blood pressure | Baseline, 16 weeks after leg heating
Change in placental growth factor level | Baseline, 16 weeks after leg heating
Change in solube fms-like tyrosine kinase-1 level | Baseline, 16 weeks after leg heating
Change in soluble endoglin level | Baseline, 16 weeks after leg heating

CONTACTS AND LOCATIONS:
Overall Officials: Qi Fu, MD, PhD, Principal Investigator — UT Southwestern Medical Center; Institute for Exercise and Environmental Medicine
Locations (1):
- UT Southwestern Medical Center; Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified individual participant data will be available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the manuscripts are published.

REFERENCES:
- [Background] Lisonkova S, Joseph KS. Incidence of preeclampsia: risk factors and outcomes associated with early- versus late-onset disease. Am J Obstet Gynecol. 2013 Dec;209(6):544.e1-544.e12. doi: 10.1016/j.ajog.2013.08.019. Epub 2013 Aug 22. PMID 23973398
- [Background] Ford ND, Cox S, Ko JY, Ouyang L, Romero L, Colarusso T, Ferre CD, Kroelinger CD, Hayes DK, Barfield WD. Hypertensive Disorders in Pregnancy and Mortality at Delivery Hospitalization - United States, 2017-2019. MMWR Morb Mortal Wkly Rep. 2022 Apr 29;71(17):585-591. doi: 10.15585/mmwr.mm7117a1. PMID 35482575
- [Background] Bicocca MJ, Mendez-Figueroa H, Chauhan SP, Sibai BM. Maternal Obesity and the Risk of Early-Onset and Late-Onset Hypertensive Disorders of Pregnancy. Obstet Gynecol. 2020 Jul;136(1):118-127. doi: 10.1097/AOG.0000000000003901. PMID 32541276
- [Background] Wang MC, Freaney PM, Perak AM, Greenland P, Lloyd-Jones DM, Grobman WA, Khan SS. Trends in Prepregnancy Obesity and Association With Adverse Pregnancy Outcomes in the United States, 2013 to 2018. J Am Heart Assoc. 2021 Sep 7;10(17):e020717. doi: 10.1161/JAHA.120.020717. Epub 2021 Aug 25. PMID 34431359
- [Background] Aksin S, Andan C, Tunc S, Goklu MR. Comparison of brachial artery flow-mediated dilatation, uterine artery Doppler, and umbilical artery Doppler measurements in obese and normal pregnant women. J Obstet Gynaecol Res. 2022 Feb;48(2):340-350. doi: 10.1111/jog.15092. Epub 2021 Nov 2. PMID 34729866
- [Background] Stewart FM, Freeman DJ, Ramsay JE, Greer IA, Caslake M, Ferrell WR. Longitudinal assessment of maternal endothelial function and markers of inflammation and placental function throughout pregnancy in lean and obese mothers. J Clin Endocrinol Metab. 2007 Mar;92(3):969-75. doi: 10.1210/jc.2006-2083. Epub 2006 Dec 27. PMID 17192290
- [Background] Petrella E, Pignatti L, Neri I, Facchinetti F. The l-arginine/nitric oxide pathway is impaired in overweight/obese pregnant women. Pregnancy Hypertens. 2014 Apr;4(2):150-5. doi: 10.1016/j.preghy.2014.01.001. Epub 2014 Feb 3. PMID 26104420
- [Background] Chin-Dusting JP, Willems L, Kaye DM. L-arginine transporters in cardiovascular disease: a novel therapeutic target. Pharmacol Ther. 2007 Dec;116(3):428-36. doi: 10.1016/j.pharmthera.2007.08.001. Epub 2007 Aug 28. PMID 17915331
- [Background] Schiffrin EL, Touyz RM. Vascular biology of endothelin. J Cardiovasc Pharmacol. 1998;32 Suppl 3:S2-13. PMID 9883741
- [Background] Schobel HP, Fischer T, Heuszer K, Geiger H, Schmieder RE. Preeclampsia -- a state of sympathetic overactivity. N Engl J Med. 1996 Nov 14;335(20):1480-5. doi: 10.1056/NEJM199611143352002. PMID 8890098
- [Background] Greenwood JP, Scott EM, Stoker JB, Walker JJ, Mary DA. Sympathetic neural mechanisms in normal and hypertensive pregnancy in humans. Circulation. 2001 Oct 30;104(18):2200-4. doi: 10.1161/hc4301.098253. PMID 11684631
- [Background] Greenwood JP, Scott EM, Walker JJ, Stoker JB, Mary DA. The magnitude of sympathetic hyperactivity in pregnancy-induced hypertension and preeclampsia. Am J Hypertens. 2003 Mar;16(3):194-9. doi: 10.1016/s0895-7061(02)03256-9. PMID 12620697
- [Background] Greenwood JP, Stoker JB, Walker JJ, Mary DA. Sympathetic nerve discharge in normal pregnancy and pregnancy-induced hypertension. J Hypertens. 1998 May;16(5):617-24. doi: 10.1097/00004872-199816050-00009. PMID 9797173
- [Background] Hissen SL, Takeda R, Badrov MB, Arias-Franklin S, Patel S, Nelson DB, Babb TG, Fu Q. Impact of maternal obesity on resting muscle sympathetic nerve activity during uncomplicated pregnancy: a longitudinal assessment. Am J Physiol Regul Integr Comp Physiol. 2024 Jan 1;326(1):R10-R18. doi: 10.1152/ajpregu.00098.2023. Epub 2023 Nov 13. PMID 37955129
- [Background] Dyakova EY, Kapilevich LV, Shylko VG, Popov SV, Anfinogenova Y. Physical exercise associated with NO production: signaling pathways and significance in health and disease. Front Cell Dev Biol. 2015 Apr 2;3:19. doi: 10.3389/fcell.2015.00019. eCollection 2015. PMID 25883934
- [Background] Wenner MM, Welti LM, Dow CA, Greiner JJ, Stauffer BL, DeSouza CA. Aerobic exercise training reduces ET-1-mediated vasoconstriction and improves endothelium-dependent vasodilation in postmenopausal women. Am J Physiol Heart Circ Physiol. 2023 Jun 1;324(6):H732-H738. doi: 10.1152/ajpheart.00674.2022. Epub 2023 Mar 24. PMID 36961490
- [Background] Maeda S, Tanabe T, Miyauchi T, Otsuki T, Sugawara J, Iemitsu M, Kuno S, Ajisaka R, Yamaguchi I, Matsuda M. Aerobic exercise training reduces plasma endothelin-1 concentration in older women. J Appl Physiol (1985). 2003 Jul;95(1):336-41. doi: 10.1152/japplphysiol.01016.2002. Epub 2003 Feb 28. PMID 12611765
- [Background] Witvrouwen I, Mannaerts D, Van Berendoncks AM, Jacquemyn Y, Van Craenenbroeck EM. The Effect of Exercise Training During Pregnancy to Improve Maternal Vascular Health: Focus on Gestational Hypertensive Disorders. Front Physiol. 2020 May 8;11:450. doi: 10.3389/fphys.2020.00450. eCollection 2020. PMID 32457655
- [Background] Boparai R, Skow RJ, Farooq S, Steinback CD, Davenport MH. Prenatal exercise and cardiovascular health (PEACH) study: the remote effect of aerobic exercise training on conduit artery and resistance vessel function. Appl Physiol Nutr Metab. 2021 Dec;46(12):1459-1468. doi: 10.1139/apnm-2020-0902. Epub 2021 Jun 23. PMID 34161737
- [Background] Skow RJ, Fraser GM, Steinback CD, Davenport MH. Prenatal Exercise and Cardiovascular Health (PEACH) Study: Impact on Muscle Sympathetic Nerve (Re)Activity. Med Sci Sports Exerc. 2021 Jun 1;53(6):1101-1113. doi: 10.1249/MSS.0000000000002583. PMID 33315812
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Background] Impact of physical activity during pregnancy and postpartum on chronic disease risk. Med Sci Sports Exerc. 2006 May;38(5):989-1006. doi: 10.1249/01.mss.0000218147.51025.8a. PMID 16672855
- [Background] Flannery C, McHugh S, Anaba AE, Clifford E, O'Riordan M, Kenny LC, McAuliffe FM, Kearney PM, Byrne M. Enablers and barriers to physical activity in overweight and obese pregnant women: an analysis informed by the theoretical domains framework and COM-B model. BMC Pregnancy Childbirth. 2018 May 21;18(1):178. doi: 10.1186/s12884-018-1816-z. PMID 29783933
- [Background] Johnson JM, Minson CT, Kellogg DL Jr. Cutaneous vasodilator and vasoconstrictor mechanisms in temperature regulation. Compr Physiol. 2014 Jan;4(1):33-89. doi: 10.1002/cphy.c130015. PMID 24692134
- [Background] Keller DM, Sander M, Stallknecht B, Crandall CG. alpha-Adrenergic vasoconstrictor responsiveness is preserved in the heated human leg. J Physiol. 2010 Oct 1;588(Pt 19):3799-808. doi: 10.1113/jphysiol.2010.194506. PMID 20693291
- [Background] Heinonen I, Brothers RM, Kemppainen J, Knuuti J, Kalliokoski KK, Crandall CG. Local heating, but not indirect whole body heating, increases human skeletal muscle blood flow. J Appl Physiol (1985). 2011 Sep;111(3):818-24. doi: 10.1152/japplphysiol.00269.2011. Epub 2011 Jun 16. PMID 21680875
- [Background] Neff D, Kuhlenhoelter AM, Lin C, Wong BJ, Motaganahalli RL, Roseguini BT. Thermotherapy reduces blood pressure and circulating endothelin-1 concentration and enhances leg blood flow in patients with symptomatic peripheral artery disease. Am J Physiol Regul Integr Comp Physiol. 2016 Aug 1;311(2):R392-400. doi: 10.1152/ajpregu.00147.2016. Epub 2016 Jun 22. PMID 27335279
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Background] Green DJ, Carter HH, Fitzsimons MG, Cable NT, Thijssen DH, Naylor LH. Obligatory role of hyperaemia and shear stress in microvascular adaptation to repeated heating in humans. J Physiol. 2010 May 1;588(Pt 9):1571-7. doi: 10.1113/jphysiol.2010.186965. Epub 2010 Mar 8. PMID 20211982
- [Background] Ely BR, Francisco MA, Halliwill JR, Bryan SD, Comrada LN, Larson EA, Brunt VE, Minson CT. Heat therapy reduces sympathetic activity and improves cardiovascular risk profile in women who are obese with polycystic ovary syndrome. Am J Physiol Regul Integr Comp Physiol. 2019 Nov 1;317(5):R630-R640. doi: 10.1152/ajpregu.00078.2019. Epub 2019 Sep 4. PMID 31483156
- [Background] Cui J, Gao Z, Leuenberger UA, Blaha C, Luck JC, Herr MD, Sinoway LI. Repeated warm water baths decrease sympathetic activity in humans. J Appl Physiol (1985). 2022 Jul 1;133(1):234-245. doi: 10.1152/japplphysiol.00684.2021. Epub 2022 Jun 23. PMID 35736952
- [Background] Naylor LH, Carter H, FitzSimons MG, Cable NT, Thijssen DH, Green DJ. Repeated increases in blood flow, independent of exercise, enhance conduit artery vasodilator function in humans. Am J Physiol Heart Circ Physiol. 2011 Feb;300(2):H664-9. doi: 10.1152/ajpheart.00985.2010. Epub 2010 Dec 3. PMID 21131471
- [Background] Tinken TM, Thijssen DH, Hopkins N, Black MA, Dawson EA, Minson CT, Newcomer SC, Laughlin MH, Cable NT, Green DJ. Impact of shear rate modulation on vascular function in humans. Hypertension. 2009 Aug;54(2):278-85. doi: 10.1161/HYPERTENSIONAHA.109.134361. Epub 2009 Jun 22. PMID 19546374
- [Background] Carter HH, Spence AL, Atkinson CL, Pugh CJ, Naylor LH, Green DJ. Repeated core temperature elevation induces conduit artery adaptation in humans. Eur J Appl Physiol. 2014 Apr;114(4):859-65. doi: 10.1007/s00421-013-2817-2. Epub 2014 Jan 8. PMID 24399113
- [Background] Laukkanen T, Khan H, Zaccardi F, Laukkanen JA. Association between sauna bathing and fatal cardiovascular and all-cause mortality events. JAMA Intern Med. 2015 Apr;175(4):542-8. doi: 10.1001/jamainternmed.2014.8187. PMID 25705824
- [Background] Patrick RP, Johnson TL. Sauna use as a lifestyle practice to extend healthspan. Exp Gerontol. 2021 Oct 15;154:111509. doi: 10.1016/j.exger.2021.111509. Epub 2021 Aug 5. PMID 34363927
- [Background] Chambers CD. Risks of hyperthermia associated with hot tub or spa use by pregnant women. Birth Defects Res A Clin Mol Teratol. 2006 Aug;76(8):569-73. doi: 10.1002/bdra.20303. PMID 16998815
- [Background] McMurray RG, Katz VL. Thermoregulation in pregnancy. Implications for exercise. Sports Med. 1990 Sep;10(3):146-58. doi: 10.2165/00007256-199010030-00002. PMID 2237032
- [Background] Ravanelli N, Casasola W, English T, Edwards KM, Jay O. Heat stress and fetal risk. Environmental limits for exercise and passive heat stress during pregnancy: a systematic review with best evidence synthesis. Br J Sports Med. 2019 Jul;53(13):799-805. doi: 10.1136/bjsports-2017-097914. Epub 2018 Mar 1. PMID 29496695
- [Background] Romero SA, Gagnon D, Adams AN, Cramer MN, Kouda K, Crandall CG. Acute limb heating improves macro- and microvascular dilator function in the leg of aged humans. Am J Physiol Heart Circ Physiol. 2017 Jan 1;312(1):H89-H97. doi: 10.1152/ajpheart.00519.2016. Epub 2016 Nov 11. PMID 27836894